CLINICAL TRIAL: NCT03079297
Title: A Pilot Double-Blind Randomized Placebo-Controlled Crossover Study to Investigate Rapid Antidepressant Effects of Leucine
Brief Title: Rapid Antidepressant Effects of Leucine
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Covid-19
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Madhukar H. Trivedi, MD, MD, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: STU 082016-037
Record Dates: First submitted 2017-03-04; First posted 2017-03-14 (Actual); Results first posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2022-12

CONDITIONS: Major Depressive Disorder
Keywords: Antidepressant; Inflammation; Biomarker; Depression; Treatment Resistant Depression; Leucine
MeSH Terms: conditions — Depressive Disorder, Major; Inflammation; Depression; Depressive Disorder, Treatment-Resistant | interventions — Leucine; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- L-leucine (Experimental): 4 gm L-leucine by mouth twice daily for two weeks
  Interventions: Drug: L-Leucine
- Maltodextrin (Placebo Comparator): 4 gm maltodextrin by mouth twice daily for two weeks
  Interventions: Other: Maltodextrin

INTERVENTIONS:
Drug: L-Leucine — L-leucine is an essential amino acid which will be provided as an effervescent powder mixture to participants.
  Other Names: Leucine
  Arms: L-leucine
Other: Maltodextrin — Maltodextrin is a nonsweet carbohydrate which will be provided as an effervescent powder mixture similar in taste and appearance to the L-leucine containing effervescent powder mixture
  Other Names: Placebo
  Arms: Maltodextrin

SUMMARY:
This randomized double-blind placebo-controlled crossover study seeks to evaluate the antidepressant effect of L-leucine, an essential amino acid, in patients with Major Depressive Disorder (MDD).

DETAILED DESCRIPTION:
This is a pilot phase II clinical trial of L-leucine to test its efficacy in reducing depressive symptoms in MDD patients, especially those who exhibit increased inflammation. The determination of increased inflammation will be done post-hoc. During the screening visit, all study participants will provide demographic information and complete self-report assessments and clinician evaluations and examinations. Blood and urine tests will also be performed. All participants who meet eligibility criteria and are willing to proceed with the study will enter this 6-week study after being randomized to two-week course of either L-leucine or placebo. In this cross-over study, participants will be crossed over to the second treatment after 2 weeks of washout. The study period will last 42 days (6 weeks) from the baseline visit. Both L-leucine and placebo will be provided as an effervescent mixture powder. Investigators hypothesize that MDD subjects will have greater reduction in depression severity on leucine as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Current primary diagnosis of nonpsychotic major depressive disorder.
* Stable antidepressant dose of no more than one antidepressant medication for 4 weeks and no anticipated changes during the study period.
* Stable doses of all concomitant medications for over 6 weeks.
* No more than two failed antidepressant trials of adequate dose and duration, as defined by ATRQ, in the current episode.

Exclusion Criteria:

* Psychiatric co-morbidity posing safety risk.
* Pregnant or breastfeeding or plan to become pregnant over the ensuing 2 months following study entry or are sexually active and not using adequate contraception
* Exclusionary psychiatric conditions (such as substance dependence in the last 6 months, substance abuse in the last 2 months, or lifetime history of psychotic disorders.
* Unstable or terminal general medical condition (GMC).
* Concomitant medications that interact with L-leucine (e.g. sildenafil).
* Vagus nerve stimulation, ECT, or rTMS, or other somatic antidepressant treatment during current episode
* Inadequately controlled hypothyroidism.
* Therapy that is depression specific, such as CBT or Interpersonal Psychotherapy of Depression.
* Hypersensitivity to L-leucine
* Have Maple Syrup Urine Disease.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2021-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhukar H Trivedi, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dantzer R, O'Connor JC, Freund GG, Johnson RW, Kelley KW. From inflammation to sickness and depression: when the immune system subjugates the brain. Nat Rev Neurosci. 2008 Jan;9(1):46-56. doi: 10.1038/nrn2297. PMID 18073775
- [Background] Jha MK, Minhajuddin A, Gadad BS, Greer T, Grannemann B, Soyombo A, Mayes TL, Rush AJ, Trivedi MH. Can C-reactive protein inform antidepressant medication selection in depressed outpatients? Findings from the CO-MED trial. Psychoneuroendocrinology. 2017 Apr;78:105-113. doi: 10.1016/j.psyneuen.2017.01.023. Epub 2017 Jan 24. PMID 28187400
- [Background] Rush AJ, Wisniewski SR, Warden D, Luther JF, Davis LL, Fava M, Nierenberg AA, Trivedi MH. Selecting among second-step antidepressant medication monotherapies: predictive value of clinical, demographic, or first-step treatment features. Arch Gen Psychiatry. 2008 Aug;65(8):870-80. doi: 10.1001/archpsyc.65.8.870. PMID 18678792
- [Background] Rush AJ, Trivedi MH, Wisniewski SR, Stewart JW, Nierenberg AA, Thase ME, Ritz L, Biggs MM, Warden D, Luther JF, Shores-Wilson K, Niederehe G, Fava M; STAR*D Study Team. Bupropion-SR, sertraline, or venlafaxine-XR after failure of SSRIs for depression. N Engl J Med. 2006 Mar 23;354(12):1231-42. doi: 10.1056/NEJMoa052963. PMID 16554525
- [Background] Trivedi MH, Fava M, Wisniewski SR, Thase ME, Quitkin F, Warden D, Ritz L, Nierenberg AA, Lebowitz BD, Biggs MM, Luther JF, Shores-Wilson K, Rush AJ; STAR*D Study Team. Medication augmentation after the failure of SSRIs for depression. N Engl J Med. 2006 Mar 23;354(12):1243-52. doi: 10.1056/NEJMoa052964. PMID 16554526

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 16 participants were consented, of which 5 were determined as eligible after screening. Of those 5, 1 reported exclusionary criteria at the baseline visit and 4 were randomized.
Groups:
- L-leucine, Then Placebo: Participants with 4 gm L-leucine by mouth twice daily for two weeks, then washout for two weeks, then 4 gm maltodextrin by mouth twice daily for two weeks.
- Placebo, Then L-leucine: Participants start with 4 gm maltodextrin by mouth twice daily for two weeks, then washout for two weeks, then 4 gm L-leucine by mouth twice daily for two weeks.
Period: First Intervention (14 Days)
Arm/Group | L-leucine, Then Placebo | Placebo, Then L-leucine
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0
Period: Washout (14 Days)
Arm/Group | L-leucine, Then Placebo | Placebo, Then L-leucine
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0
Period: Second Intervention (14 Days)
Arm/Group | L-leucine, Then Placebo | Placebo, Then L-leucine
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- A/B (L-leucine/Maltodextrin): Starts with 4 gm L-leucine by mouth twice daily for two weeks, then washout for two weeks, then 4 gm maltodextrin by mouth twice daily for two weeks.
- B/A (Maltodextrin/L-leucine): Starts with 4 gm maltodextrin by mouth twice daily for two weeks, then washout for two weeks, then 4 gm L-leucine by mouth twice daily for two weeks.
- Total: Total of all reporting groups
Arm/Group | A/B (L-leucine/Maltodextrin) | B/A (Maltodextrin/L-leucine) | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in QIDS-SR From Baseline at 14 Days
Description: The Quick Inventory of Depressive Symptomatology, self-report (QIDS-SR), self-report is a 16-item measure of depression severity that includes the 9 criterion symptoms for MDD. Items are scored on a 4-point Likert scale, ranging from 0 to 3 (total score range, 0-27). Totals scores of ≤ 5 indicate no depression; 6-10 indicates mild depression; 11-15 indicates moderate depression; 16-20 indicates severe depression; and ≥ 21 indicates very severe depression. For purposes of this report, severe and very severe categories were combined as "severe to very severe" depression (≥ 16). The QIDS-A self-report has demonstrated acceptable psychometric properties.
Time Frame: Baseline to 14 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | L-leucine | Maltodextrin
Number analyzed (Participants) | 4 | 4
score on a scale | -6 (3.16) | -8 (3.27)
Statistical Analysis 1: Comparison: L-leucine vs Maltodextrin; Test type: Superiority; p = 0.4128, t-test, 2 sided; Mean Difference (Final Values) = 2, 95% CI 2-sided [-3.56 to 7.56], Standard Error of Mean 2.5000

2. Secondary Outcome: Percentage of MDD Patients With 50% or Greater Reduction in Depression Severity After 14 Days of LEU and PBO Treatments.
Description: Response criteria defined based on QIDS-SR score at baseline and 14 days after treatment initiation.
  The Quick Inventory of Depressive Symptomatology, self-report (QIDS-SR), self-report is a 16-item measure of depression severity that includes the 9 criterion symptoms for MDD. Items are scored on a 4-point Likert scale, ranging from 0 to 3 (total score range, 0-27). Totals scores of ≤ 5 indicate no depression; 6-10 indicates mild depression; 11-15 indicates moderate depression; 16-20 indicates severe depression; and ≥ 21 indicates very severe depression. For purposes of this report, severe and very severe categories were combined as "severe to very severe" depression (≥ 16). The QIDS-A self-report has demonstrated acceptable psychometric properties.
Time Frame: Baseline to 14 days
Measure: Number; unit: percentage of patients
Arm/Group | L-leucine | Maltodextrin
Number analyzed (Participants) | 4 | 4
percentage of patients | 0 | 50
Statistical Analysis 1: Comparison: L-leucine; Test type: Superiority; p = 0.4286, Fisher Exact

3. Secondary Outcome: Percentage of MDD Patients With QIDS-SR Score Less Than or Equal to 5 at 14 Days of LEU and PBO Treatments.
Description: Remission operationalized as QIDS-SR <=5.
  The Quick Inventory of Depressive Symptomatology, self-report (QIDS-SR), self-report is a 16-item measure of depression severity that includes the 9 criterion symptoms for MDD. Items are scored on a 4-point Likert scale, ranging from 0 to 3 (total score range, 0-27). Totals scores of ≤ 5 indicate no depression; 6-10 indicates mild depression; 11-15 indicates moderate depression; 16-20 indicates severe depression; and ≥ 21 indicates very severe depression. For purposes of this report, severe and very severe categories were combined as "severe to very severe" depression (≥ 16). The QIDS-A self-report has demonstrated acceptable psychometric properties.
Time Frame: 14 days
Measure: Number; unit: percentage of patients
Arm/Group | L-leucine | Maltodextrin
Number analyzed (Participants) | 4 | 4
percentage of patients | 0 | 25
Statistical Analysis 1: Comparison: L-leucine vs Maltodextrin; Test type: Superiority; p = .999, Fisher Exact

4. Secondary Outcome: Rates of Adverse Effects After 3 Days, 7 Days and 14 Days of LEU and PBO Treatments.
Description: Adverse effect burden will be measured with Frequency Intensity and Burden of Side-effect rating scale (FIBSER).
  The Frequency, Intensity, Burden of Side Effects Rating (FIBSER) scale was designed by Dr. Stephen Wisniewski for use in the U.S. STAR*D effectiveness study. It is a 3-item scale to assess side effects from antidepressant treatment. To use the FIBSER in measurement-based care, clinicians should consider item 3 (Burden). If the score is 0 to 2 (None to Mild interference with activities), no change in medication is needed. If the score is 3-4 (Moderate to Marked interference with activites), the side effects need to be addressed (i.e., change in dose, side effect antidote, etc). If the score is 5-6 (Severe interference with activities or Unable to Function), the dose needs to be decreased or the medication needs to be switched.
Time Frame: Baseline to 3 days, 7 days, and 14 days
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | L-leucine | Maltodextrin
Number analyzed (Participants) | 4 | 4
units on a scale
  Adverse effect burden 3 days Change | 0 (.07) | 0 (.06)
  Adverse effect burden function 7 days Change | 0 (.07) | 0 (.06)
  Adverse effect burden function 14 days Change | 0 (.06) | -.25 (.06)
Statistical Analysis 1: Comparison: L-leucine vs Maltodextrin; Test type: Superiority; p = 0.9932, MMRM — P-value for Adverse effect burden 3 days Change. Model: Change from baseline=Baseline, Visit, Treatment, Treatment*Visit
Statistical Analysis 2: Comparison: L-leucine vs Maltodextrin; Test type: Superiority; p = 0.9932, MMRM — P-value for Adverse effect burden 7 days Change. Model: Change from baseline=Baseline, Visit, Treatment, Treatment*Visit
Statistical Analysis 3: Comparison: L-leucine vs Maltodextrin; Test type: Superiority; p = 0.2242, MMRM — P-value for Adverse effect burden 14 days Change. Model: Change from baseline=Baseline, Visit, Treatment, Treatment*Visit

5. Secondary Outcome: Change in Fatigue Symptoms From Baseline After 3, 7, and 14 Days of LEU and PBO Treatments Measured With Multidimensional Fatigue Inventory.
Description: Fatigue will be measured with Multidimensional fatigue inventory
  The Multidimensional Fatigue Inventory (MFI) is a 20-item self-report instrument designed to measure fatigue. It contains five scales: general fatigue (items 1, 5, 12, 16), mental fatigue (items 7, 11, 13, 19), physical fatigue (items 2, 8, 14, 20), reduced motivation (items 4, 9, 15, 18) and reduced activity (items 3, 6, 10, 17). Items are scored on a 5-point scale on which the participant expressed the degree to which the statement applied to him or her (from agreement "yes, that is true" to disagreement "no, that is not true") in the previous days. Item scores are summed to create a sum score for each scale, ranging between 4 (best condition) and 20 (worst condition). Higher scores indicate more fatigue.
Time Frame: Baseline to 3 days, 7 days, and 14 days
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | L-leucine | Maltodextrin
Number analyzed (Participants) | 4 | 4
units on a scale
  General fatigue 3 days Change | -1.59 (1.93) | -0.70 (1.66)
  General fatigue 7 days Change | -3.59 (1.93) | -3.20 (1.66)
  General fatigue 14 days Change | -0.74 (1.67) | -3.70 (1.66)
  Mental fatigue 3 days Change | -2.36 (1.71) | -0.71 (1.62)
  Mental fatigue 7 days Change | -1.02 (1.71) | -4.71 (1.62)
  Mental fatigue 14 days Change | -3.46 (1.62) | -3.96 (1.62)
  Physical fatigue 3 days Change | -3.58 (1.16) | -0.55 (1.08)
  Physical fatigue 7 days Change | 0.09 (1.16) | -1.80 (1.08)
  Physical fatigue 14 days Change | -2.55 (1.08) | -3.80 (1.08)
  Reduced motivation 3 days Change | -.032 (1.72) | -0.26 (1.59)
  Reduced motivation 7 days Change | -0.71 (1.94) | -1.26 (1.59)
  Reduced motivation 14 days Change | -5.51 (1.59) | -2.76 (1.59)
  Reduced activity 3 days Change | -2.80 (1.68) | -0.47 (1.51)
  Reduced activity 7 days Change | -4.14 (1.68) | -3.97 (1.51)
  Reduced activity 14 days Change | -4.47 (1.51) | -8.14 (1.68)
Statistical Analysis 1: Comparison: L-leucine vs Maltodextrin; Test type: Superiority; p = 0.7282, MMRM — P-value for General fatigue 3 days Change. Model: Change from baseline=Baseline, Visit, Treatment, Treatment*Visit
Statistical Analysis 2: Comparison: L-leucine vs Maltodextrin; Test type: Superiority; p = 0.8781, MMRM — P-value for General fatigue 7 days Change. Model: Change from baseline=Baseline, Visit, Treatment, Treatment*Visit
Statistical Analysis 3: Comparison: L-leucine vs Maltodextrin; Test type: Superiority; p = 0.226, MMRM — P-value for General fatigue 14 days Change. Model: Change from baseline=Baseline, Visit, Treatment, Treatment*Visit
Statistical Analysis 4: Comparison: L-leucine vs Maltodextrin; Test type: Superiority; p = 0.2158, MMRM — P-value for Mental fatigue 3 days Change. Model: Change from baseline=Baseline, Visit, Treatment, Treatment*Visit
Statistical Analysis 5: Comparison: L-leucine vs Maltodextrin; Test type: Superiority; p = 0.0081, MMRM — P-value for Mental fatigue 7 days Change. Model: Change from baseline=Baseline, Visit, Treatment, Treatment*Visit
Statistical Analysis 6: Comparison: L-leucine vs Maltodextrin; Test type: Superiority; p = 0.6768, MMRM — P-value for Mental fatigue 14 days Change. Model: Change from baseline=Baseline, Visit, Treatment, Treatment*Visit
Statistical Analysis 7: Comparison: L-leucine vs Maltodextrin; Test type: Superiority; p = 0.0076, MMRM — P-value for Physical fatigue 3 days Change. Model: Change from baseline=Baseline, Visit, Treatment, Treatment*Visit
Statistical Analysis 8: Comparison: L-leucine vs Maltodextrin; Test type: Superiority; p = 0.0858, MMRM — P-value for Physical fatigue 7 days Change. Model: Change from baseline=Baseline, Visit, Treatment, Treatment*Visit
Statistical Analysis 9: Comparison: L-leucine vs Maltodextrin; Test type: Superiority; p = 0.2065, MMRM — P-value for Physical fatigue 14 days Change. Model: Change from baseline=Baseline, Visit, Treatment, Treatment*Visit
Statistical Analysis 10: Comparison: L-leucine vs Maltodextrin; Test type: Superiority; p = 0.9712, MMRM — P-value for Reduced motivation 3 days Change. Model: Change from baseline=Baseline, Visit, Treatment, Treatment*Visit
Statistical Analysis 11: Comparison: L-leucine vs Maltodextrin; Test type: Superiority; p = 0.7572, MMRM — P-value for Reduced motivation 7 days Change. Model: Change from baseline=Baseline, Visit, Treatment, Treatment*Visit
Statistical Analysis 12: Comparison: L-leucine vs Maltodextrin; Test type: Superiority; p = 0.0588, MMRM — P-value for Reduced motivation 14 days Change. Model: Change from baseline=Baseline, Visit, Treatment, Treatment*Visit
Statistical Analysis 13: Comparison: L-leucine vs Maltodextrin; Test type: Superiority; p = 0.1857, MMRM — P-value for Reduced activity 3 days Change. Model: Change from baseline=Baseline, Visit, Treatment, Treatment*Visit
Statistical Analysis 14: Comparison: L-leucine vs Maltodextrin; Test type: Superiority; p = 0.9225, MMRM — P-value for Reduced activity 7 days Change. Model: Change from baseline=Baseline, Visit, Treatment, Treatment*Visit
Statistical Analysis 15: Comparison: L-leucine vs Maltodextrin; Test type: Superiority; p = 0.0414, MMRM — P-value for Reduced activity 14 days Change. Model: Change from baseline=Baseline, Visit, Treatment, Treatment*Visit

6. Secondary Outcome: Change in Psychosocial Function From Baseline After 3, 7, and 14 Days of LEU and PBO Treatments Measured Using Work and Social Adjustment Scale.
Description: Psychosocial function will be measured using Work and Social Adjustment Scale
  The Work and Social Adjustment Scale ("WSAS") is a 5-item measure for impairment in functioning. Items are scored on an 8-point scale on how much participants' problems impaired their ability to carry out the activity (from "Not at all" to "Very severely"). Item scores are summed to create a sum score. The maximum score of the WSAS is 40, lower scores are better. A WSAS score above 20 appears to suggest moderately severe or worse psychopathology. Scores between 10 and 20 are associated with significant functional impairment but less severe clinical symptomatology. Scores below 10 appear to be associated with subclinical populations.
Time Frame: Baseline to 3 days, 7 days, and 14 days
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | L-leucine | Maltodextrin
Number analyzed (Participants) | 4 | 4
units on a scale
  Psychosocial function 3 days Change | 1.49 (5.14) | -2.57 (4.44)
  Psychosocial function7 days Change | -1.18 (5.14) | -7.57 (4.44)
  Psychosocial function 14 days Change | -9.38 (4.46) | -7.32 (4.44)
Statistical Analysis 1: Comparison: L-leucine vs Maltodextrin; Test type: Superiority; p = 0.4603, MMRM — P-value for Psychosocial function 3 days Change. Model: Change from baseline=Baseline, Visit, Treatment, Treatment*Visit
Statistical Analysis 2: Comparison: L-leucine vs Maltodextrin; Test type: Superiority; p = 0.2521, MMRM — P-value for Psychosocial function 7 days Change. Model: Change from baseline=Baseline, Visit, Treatment, Treatment*Visit
Statistical Analysis 3: Comparison: L-leucine vs Maltodextrin; Test type: Superiority; p = 0.6635, MMRM — P-value for Psychosocial function 14 days Change. Model: Change from baseline=Baseline, Visit, Treatment, Treatment*Visit

7. Secondary Outcome: Change in Anhedonia From Baseline After 3, 7, and 14 Days of LEU and PBO Treatments Measured Using Snaith-Hamilton Pleasure Scale (SHAPS)
Description: Anhedonia will be measured using Snaith-Hamilton Pleasure Scale (SHAPS).
  The Snaith-Hamilton Pleasure Scale (SHAPS) is a 14-item scale that measures anhedonia, the inability to experience pleasure. The items cover the domains of: social interaction, food and drink, sensory experience, and interest/pastimes. A score of 2 or less constitutes a "normal" score, while an "abnormal" score is defined as 3 or more. Each item has four possible responses: strongly disagree, disagree, agree, or strongly agree. Either of the "disagree" responses score one point, and either of the "agree" responses score 0 points. Thus, the final score ranges from 0 to 14.
Time Frame: Baseline to 3 days, 7 days, and 14 days
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | L-leucine | Maltodextrin
Number analyzed (Participants) | 4 | 4
units on a scale
  Anhedonia 3 days Change | -0.21 (0.75) | -0.46 (0.65)
  Anhedonia 7 days Change | 0.79 (0.75) | -1.46 (0.65)
  Anhedonia 14 days Change | -0.07 (0.66) | -2.21 (0.65)
Statistical Analysis 1: Comparison: L-leucine vs Maltodextrin; Test type: Superiority; p = 0.7839, MMRM — P-value for Anhedonia 3 days Change. Model: Change from baseline=Baseline, Visit, Treatment, Treatment*Visit
Statistical Analysis 2: Comparison: L-leucine vs Maltodextrin; Test type: Superiority; p = 0.0248, MMRM — P-value for Anhedonia function 7 days Change. Model: Change from baseline=Baseline, Visit, Treatment, Treatment*Visit
Statistical Analysis 3: Comparison: L-leucine vs Maltodextrin; Test type: Superiority; p = 0.0199, MMRM — P-value for Anhedonia 14 days Change. Model: Change from baseline=Baseline, Visit, Treatment, Treatment*Visit

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected for each participant from their Baseline Visit (Day 0) to Day 42, for a total of 43 days.
Description: Adverse events were assessed at the end of each visit.
Groups:
- L-leucine: AE was reported with a start date within the two week period subject was taking 4 gm L-leucine by mouth twice daily
- Washout Following L-Leucine: AE was reported with a start date following (within two weeks) the two week period subject was taking 4 gm L-leucine by mouth twice daily
- Maltodextrin: AE was reported with a start date within the two week period subject was taking 4 gm Maltodextrin by mouth twice daily
- Washout Following Maltodextrin: AE was reported with a start date following (within two weeks) the two week period subject was taking 4 gm Maltodextrin by mouth twice daily
Arm/Group | L-leucine | Washout Following L-Leucine | Maltodextrin | Washout Following Maltodextrin
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 1/4 | 1/4 | 2/4 | 2/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L-leucine (N=4) | Washout Following L-Leucine (N=4) | Maltodextrin (N=4) | Washout Following Maltodextrin (N=4)
Neutrophil count low (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
White blood cell count low (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AST Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Red blood cell count low (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemoglobin low (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematocrit low (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mean cell hemoglobin concentration increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count low (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Monocyte count low (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-16): https://cdn.clinicaltrials.gov/large-docs/97/NCT03079297/Prot_SAP_000.pdf